CLINICAL TRIAL: NCT03134248
Title: Bilateral Dispensing Study of MyDay Toric, 1-day Acuvue Moist for Astigmatism, and Dailies Aquacomfort Plus Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-72
Record Dates: First submitted 2017-04-12; First posted 2017-04-28 (Actual); Results first posted 2018-06-26 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- MyDay Toric (Experimental): Participants were randomized to wear a new pair of MyDay Toric lenses each day for one week during the cross over study
  Interventions: Device: MyDay Toric
- 1-Day Acuvue Moist for Astigmatism (Active Comparator): Participants were randomized to wear a new pair of 1-Day Acuvue Moist Toric lenses each day for one week during the cross over study
  Interventions: Device: 1-Day Acuvue Moist for Astigmatism
- Dailies Aquacomfort Plus Toric (Active Comparator): Participants were randomized to wear a new pair of Dailies Aquacomfort Plus Toric lenses each day for one week during the cross over study
  Interventions: Device: Dailies Aquacomfort Plus Toric

INTERVENTIONS:
Device: Dailies Aquacomfort Plus Toric — daily disposable contact lens
  Other Names: DACP
  Arms: Dailies Aquacomfort Plus Toric
Device: 1-Day Acuvue Moist for Astigmatism — daily disposable contact lens
  Other Names: 1-Day AM
  Arms: 1-Day Acuvue Moist for Astigmatism
Device: MyDay Toric — daily disposable contact lens
  Other Names: MDT
  Arms: MyDay Toric

SUMMARY:
Bilateral dispensing study of MyDay Toric, 1-day Acuvue Moist for Astigmatism, and Dailies Aquacomfort Plus Toric lenses

DETAILED DESCRIPTION:
Prospective, double-masked (investigator and participant), bilateral, randomized, cross-over dispensing study comparing the MyDay Toric (test) against the 1-day Acuvue Moist for Astigmatism (control), and Dailies Aquacomfort Plus Toric (control) lenses

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has had a self-reported oculo-visual examination in the last two years.
3. Has read and signed an information consent letter;
4. Is willing and able to follow instructions and maintain the appointment schedule;
5. Is an adapted soft contact lens wearer;
6. Is willing to wear contact lens in both eyes for the duration of the study;
7. Has a minimum spectacle astigmatism of - 0.75;
8. Can be fit with the three study contact lens types in the powers available;
9. Has a visual acuity of 20/30 or better in each eye with habitual correction, or 20/20 best corrected vision (for binocular distance acuity);
10. Can achieve a distance visual acuity of 20/30 (0.18 logMar) or better in each eye with the study contact lenses.
11. Has clear corneas and no active* ocular disease;

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Exclusion Criteria:

1. Is participating in any concurrent clinical trial;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to fluorescein dye or products to be used in the study;
6. Appears to have any active* ocular pathology, ocular anomaly or severe insufficiency of lacrimal secretion (severe dry eye) that would affect the wearing of contact lenses;
7. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
8. Is aphakic;
9. Has undergone refractive error surgery.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CCLR, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 subjects were enrolled for this study (assigned a subjectID), but 11 of these subjects were screen failures, leaving 49 subjects who were randomized for lens assignments.
Groups:
- 1-Day AM First, Then DACP, Then MDT: 1-day Acuvue Moist for Astig first, then Dailies Aquacomfort Plus, then MyDay Troic
- 1-Day AM First, Then MDT, Then DACP: 1-day Acuvue Moist for Astig, then MyDay Toric, then Dailies Aquacomfort Plus
- DACP First, Then 1-Day AM, Then MDT: Dailies Aquacomfort Plus, then 1-day Acuvue Moist for Astig, then MyDay Toric
- DACP First, Then MDT, Then 1-Day AM: Dailies Aquacomfort Plus, then MyDay Toric, then 1-day Acuvue Moist for Astig
- MDT First, Then 1-Day AM, Then DACP: MyDay Toric, then 1-day Acuvue Moist for Astig, then Dailies Aquacomfort Plus
- MDT First, Then DACP, Then 1-Day AM: MyDay Toric, then Dailies Aquacomfort Plus, then 1-day Acuvue Moist for Astig
Period: Week 1
Arm/Group | 1-Day AM First, Then DACP, Then MDT | 1-Day AM First, Then MDT, Then DACP | DACP First, Then 1-Day AM, Then MDT | DACP First, Then MDT, Then 1-Day AM | MDT First, Then 1-Day AM, Then DACP | MDT First, Then DACP, Then 1-Day AM
Started | 7 | 8 | 9 | 7 | 9 | 9
Completed | 7 | 8 | 9 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 2
Arm/Group | 1-Day AM First, Then DACP, Then MDT | 1-Day AM First, Then MDT, Then DACP | DACP First, Then 1-Day AM, Then MDT | DACP First, Then MDT, Then 1-Day AM | MDT First, Then 1-Day AM, Then DACP | MDT First, Then DACP, Then 1-Day AM
Started | 7 | 8 | 9 | 7 | 9 | 9
Completed | 7 | 8 | 9 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 3
Arm/Group | 1-Day AM First, Then DACP, Then MDT | 1-Day AM First, Then MDT, Then DACP | DACP First, Then 1-Day AM, Then MDT | DACP First, Then MDT, Then 1-Day AM | MDT First, Then 1-Day AM, Then DACP | MDT First, Then DACP, Then 1-Day AM
Started | 7 | 8 | 9 | 7 | 9 | 9
Completed | 7 | 8 | 9 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: A bilateral dispensing of MyDay Toric, 1-Day Acuvue Moist for Astigmatism, and Dailies Aqua Comfort Plus Toric Contact Lenses
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 49

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings of lens performance for comfort assessed. Comfort Scale 0-10, 0=painful, 10=can't feel the lenses.
Time Frame: 1 week
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- MyDay Toric Contact Lens: Participants randomly assigned to wear MyDay Toric lenses either as first, second or third lens in this crossover study.
- 1-Day Acuvue Moist for Astigmatism Contact Lens: Participants randomly assigned to wear 1-Day Acuvue Moist for Astigmatism contact lenses either as first, second or third lens in this crossover study.
- Dailies Aquacomfort Plus Toric Contact Lens: Participants randomly assigned to wear Dailies Aquacomfort Plus Toric lenses either as first, second or third lens in this crossover study.
Arm/Group | MyDay Toric Contact Lens | 1-Day Acuvue Moist for Astigmatism Contact Lens | Dailies Aquacomfort Plus Toric Contact Lens
Number analyzed (Participants) | 49 | 49 | 49
units on a scale | 8 (1.37) | 9 (1.14) | 8 (2.05)

2. Primary Outcome: Dryness
Description: Subjective ratings of lens performance for dryness assessed. Dryness Scale 0-10, 0=extremely dry, 10=no dryness
Time Frame: 1 week
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | MyDay Toric Contact Lens | 1-Day Acuvue Moist for Astigmatism Contact Lens | Dailies Aquacomfort Plus Toric Contact Lens
Number analyzed (Participants) | 49 | 49 | 49
units on a scale | 9 (1.69) | 8 (1.65) | 7 (2.18)

3. Primary Outcome: Visual Quality
Description: Subjective ratings of lens performance for visual quality assessed. Visual quality Scale 0-10, 0=completely dissatisfied, 10=completely satisfied
Time Frame: 1 week
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | MyDay Toric Contact Lens | 1-Day Acuvue Moist for Astigmatism Contact Lens | Dailies Aquacomfort Plus Toric Contact Lens
Number analyzed (Participants) | 49 | 49 | 49
units on a scale | 9 (1.41) | 8 (1.14) | 8 (1.81)

4. Primary Outcome: Lens Preference With Respect to Overall Comfort
Description: Overall comfort preference of MyDay Toric, 1-Day Acuvue Moist Toric or Dailies Aquacomfort Plus Toric lenses. Scale: Strong or Slight preference for one lens, or No-preference
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Overall comfort preference of MyDay Toric, 1-Day Acuvue Moist Toric or Dailies Aquacomfort Plus Toric lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 49
Participants
  Strongly Prefer MyDay Toric | 15
  Slightly Prefer MyDay Toric | 6
  Strongly Prefer 1Day Acuvue Moist Toric | 14
  Slightly Prefer 1Day Acuvue Moist Toric | 5
  Strongly Prefer Dailies Aquacomfort Plus Toric | 5
  Slighlty Prefer Dailies Aquacomfort Plus Toric | 3
  No Preference | 1

5. Primary Outcome: Lens Preference With Respect to Visual Quality
Description: Overall visual quality preference of MyDay Toric, 1-Day Acuvue Moist Toric or Dailies Aquacomfort Plus Toric lenses. Scale: Strong or Slight preference for one lens, or No-preference
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: A bilateral dispensing of MyDay Toric, 1-Day Acuvue Moist for Astigmatism, and Dailies Aqua Comfort Plus Toric Lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 49
Participants
  Strongly Prefer MyDay Toric | 10
  Slightly Prefer MyDay Toric | 4
  Strongly Prefer 1Day Acuvue Moist Toric | 9
  Slightly Prefer 1Day Acuvue Moist Toric | 8
  Strongly Prefer Dailies Aquacomfort Plus Toric | 6
  Slightly Prefer Dailies Aquacomfort Plus Toric | 2
  No Preference | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 3 week study duration.
Description: Adverse event information was routinely collected during the weekly visits over the study duration or self-reported by the subjects if event was realized outside of visits.
Groups:
- MyDay Toric: Participants who wore MyDay Toric contact lenses
- 1-Day Acuvue Moist for Astigmatism: Participants who wore 1-Day Acuvue Moist for Astigmatism contact lenses
- Dailies Aqua Comfort Plus Toric: Participants who wore Dailies Aqua Comfort Plus Toric contact lenses
Arm/Group | MyDay Toric | 1-Day Acuvue Moist for Astigmatism | Dailies Aqua Comfort Plus Toric
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03134248/Prot_SAP_001.pdf